CLINICAL TRIAL: NCT04262622
Title: Postoperative Analgesia for Elective Mid-line Laparotomies: Thoracic Epidural Versus Surgically-placed Rectus Sheath Catheters
Brief Title: Analgesia for Mid-line Laparotomies: Thoracic Epidural vs Restus Sheath Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Salwa Hassan Waly, Associate Professor of Anesthesia and Surgical Intensive Care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5902-22-5-2019
Record Dates: First submitted 2020-01-27; First posted 2020-02-10 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Mid-line Laparotomies
Keywords: thoracic epidural analgesia; rectus sheath block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TEA (Active Comparator)
  Interventions: Device: Group RSB: rectus sheath block group
- Group RSB (Active Comparator)
  Interventions: Device: Group TEA: thoracic epidural analgesia group

INTERVENTIONS:
Device: Group TEA: thoracic epidural analgesia group — in this group TEA will be performed by the insertion of transthoracic epidural catheter before induction of general anesthesia. Analgesia will be started on wound closure by injecting local anesthetic mixture into the epidural catheter
  Arms: Group RSB
Device: Group RSB: rectus sheath block group — Two sets of epidural catheters which have multiple perforations at the end of the tubing will be surgically applied bilaterally into the rectus sheaths for each patient in this group on wound closure. By the end of surgery,injection of local anesthetic mixture will be started.
  Arms: Group TEA

SUMMARY:
Midline laparotomies are accompanied by severe postoperative pain. Adequate post-operative pain relief after major abdominal surgery reduces complications (e.g. chest infection or deep venous thrombosis) and enhances recovery and early mobilization, with better patients' satisfaction, and less hospital stay.

The standard technique for post-operative analgesia after major abdominal surgery is thoracic epidural analgesia (TEA). On the other hand, the complications encountered with TEA motivates the search for another technique, besides that in some situations, midline incision is needed while TEA is contraindicated e.g. emergency laparotomy.

Rectus sheath nerve block (RSB) is a regional anesthetic technique that provides midline somatic analgesia and might be an alternative to TEA. It is an old technique that has been revisited because of the availability of new local anesthetic agents, and the availability of small-caliber catheters.

It was hypothesized that rectus sheath analgesia (RSA) might be an alternative to thoracic epidural analgesia. Thereby, the aim of the current study is to find whether analgesia provided through surgically placed rectus sheath catheters can be a safe and effective alternative to thoracic epidural analgesia for postoperative pain relief in patients undergoing elective midline laparotomies.

DETAILED DESCRIPTION:
Administrative design:

* Approval is obtained from the ethics committee of faculty of medicine, IRB approval and the Department of Anesthesia and Surgical Intensive Care, Zagazig University.
* Informed written consent will be obtained from all patients in the study.
* The patient has the right to withdraw from the study at any time without negative sequences on their medical or surgical treatment plan.

Sample size:

The power of this study is calculated prospectively using G*POWER program version 3.1.9.2. (Heinrich Heine; Universitat Dusseldorf; Germany). To calculate sample size, degree of postoperative analgesia is used as the primary outcome. A pilot study (10 patients in each group) was performed to detect significant difference in the degree of postoperative analgesia (following VAS). It is found that 24 patients are needed in each group to achieve an alpha error level of 0.05, with 80% power and 95% confidence interval. Allowing a 5% drop out rate, the final sample size needed is 25 patients in each group to detect clinically significant difference of >20%.

Statistical analysis plan Categorical data will be presented as frequencies and/or percentages and analyzed with a chi-square or Fisher's exact test. Quantitative variables will be analyzed with unpaired t test. Statistical analysis will be performed using IBM SPSS Statistics (version 21). A p value equal to or less than 0.05 was considered statistically significant.

Study Design:

Patients will be randomly assigned to one of two groups using computer generated randomization tables:

• Thoracic epidural analgesia group (Group TEA): The skin and subcutaneous tissues will be infiltrated using 1 mL lidocaine 2% approximately lateral to the inferior aspect of the targeted spinous process using a 1.5-inch 25-gauge needle. A 17-gauge Tuohy needle will be introduced through paramedian approach. For all patients in this group, the needle will be introduced at T7 to T9. A test dose of 3 mL of lidocaine 2% with 1:200,000 adrenaline will be injected through the epidural catheter followed by induction of general anesthesia. On wound closure 20 mL 0.25% bupivacaine + 40 μg Fentanyl will be injected into the epidural catheter. Thereafter, in post-anesthesia care unit (PACU) and in surgical intensive care unit (SICU), 20 mL of 0.125% bupivacaine + 40 μg Fentanyl will be administered every 6 h for 48 hours.

• Rectus sheath block group (Group RSB): Touhy needle will be inserted 2-4 cm lateral to the midline in an angle of 45 degrees to the skin, through the anterior abdominal wall until reaching the potential space between the posterior layer of the rectus sheath and rectus abdominis muscle. The catheter will be surgically inserted into the rectus sheath. The surgeon will put the nondominant hand inside the abdomen to locate the needle tip and the other hand gently push the epidural needle in the interface between the peritoneum and muscle layer. The catheters will be placed at the upper end of the laparotomy wound until a 5cm length is inside the rectus sheath. After securing the catheter, it will be flushed with saline 0.9% and the same procedure will be repeated on the other side. After that 20 mL of 0.125% bupivacaine + 20 μg Fentanyl will be injected in each catheter as an initial bolus dose to block the intercostal nerves to provide analgesia through the recovery period until the next dose. In PACU and in SICU, 10 mL of 0.125% bupivacaine + 20 μg Fentanyl every 6 hours will be administered into each catheter for 48 hours.

Patients' monitoring and general anesthesia for both groups All patients will be closely monitored with electrocardiography, pulse oximetry, sphygmomanometer cuff and capnography. Anesthesia will be induced by 1 µg/kg fentanyl, propofol 2 mg/kg slowly, and rocuronium bromide at a dose of 0.5 mg/kg to facilitate endotracheal tube insertion. Following induction, mechanical ventilation of the lungs will be applied to maintain end tidal carbon dioxide between 35-40 mmHg. Anesthesia will be maintained using 1.5 MAC isoflurane. Subsequent doses of rocuronium 0.01 mg/kg will be given if needed (according to nerve stimulator train of four (TOF) response). Additional doses of fentanyl 1 µg/kg will be given following clinical data of the patient (if both heart rate and mean arterial blood pressure increases >20% from baseline despite maintaining adequate depth of anesthesia). By the end of surgery, reversal of neuromuscular block will be performed using neostigmine 0.05 mg/kg and atropine 0.02 mg/kg and patients will be extubated before transfer to PACU.

• For both groups: IV 1 gm paracetamol (Perfalgan)/ 8h will be given to patients. The first dose of paracetamol will be given intraoperatively on wound closure.

Opioid-based patient-driven titration protocols have been previously applied in other studies [19, 20]. Thereby, for patients in both groups, if breakthrough pain occurred, the following plan will be applied: ensure that the analgesic protocol of the study is followed then evaluate the degree of pain according to visual analogue scale (VAS) [1] where 0= no pain, and 10= worst pain possible. If VAS is ≥4= inadequate pain relief, Fentanyl-based patient-driven titration protocol will be followed for supplementary IV analgesia: the patient will be given 25 µg fentanyl, if after 5 min VAS is still ≥ 4, another 25µg fentanyl will be given, to be repeated every 5 min if needed with a maximum dose of 1 µg/kg of fentanyl.

Failure of the intervention is defined as complete absence of sensory blockade with no improvement in pain severity as reported by the patient after an adequate bolus injection of local anesthetic through either the TEA or RSC. Cases will be recorded if occurred.

Data collection:

Baseline data will be collected from all patients during a visit 24 hours before surgery. From all patients, the following data will be collected during intra- and post-operative periods (for 48 hours) as follows:

1. Vital signs [including Mean arterial blood pressure (MAP), Heart rate (HR), and Respiratory rate (RR)] will be recorded every 10 min during intraoperative period. During postoperative period, they will be recorded every 10 min for the first hour after each time of administration of local anesthetic into the catheters. For the next 5 hours, they will be recorded every one hour. This process will be repeated during the first 48 h of post-operative period.
2. Patient oxygenation will be recorded during intraoperative period and the first 48h of post-operative period.
3. Degree of postoperative pain (using VAS score) [1] and sedation level (using Ramsay sedation scale (RSS) [2], will be evaluated and recorded at the following postoperative times: 0, 3, 6, 12, 24, 36 and 48 hours; where T0= time of arrival of the patient to PACU.
4. Time to first dose of supplementary analgesia with IV Fentanyl will be recorded in each group (starting from the time of administration of the first dose of local anesthetic into the catheters, to time of VAS ≥ 4).
5. Total intra- and post-operative consumption of Fentanyl in each group.
6. Complications will be recorded and managed if occurred.
7. After discharge from operation room, all patients will be monitored at 1-hour intervals for the presence of bowel sounds and/or the passage of flatus in order to allow oral fluid intake. Time of initiation of oral fluid intake will be recorded in both groups. Times for the patient to be able to ambulate independently will be also recorded. The starting time-point for both functions will be the time of administration of the first dose of local anesthetic into the catheters, while the end-point will be the time when the patient will be able to perform these functions).
8. Patient satisfaction regarding postoperative pain control using a scale of 1-3 (3-Good, 2-Fair, 1-Poor) will be recorded.

Results Collected data will be presented in tables and/or suitable graphs and analyzed by computer software (SPSS statistics) using appropriate statistical methods and will be compared to relevant literatures and scientific researches.

ELIGIBILITY:
Inclusion Criteria:

1. Patient acceptance.
2. American Society of Anesthesiology (ASA) physical status classification of I - III
3. Body mass index (BMI) of 18.5-29.9 kg/m2
4. Patients who are posted for elective abdominal operations with midline incision under general anesthesia (e.g. colorectal resections including right or left hemicolectomy or segmental colonic resection).

Exclusion Criteria:

1. Extensive surgery beyond midline incision (e.g. abdomino-perineal resection)
2. Coagulopathies.
3. Local infection at sites of catheters insertion.
4. Systemic sepsis.
5. Severe cardiac or respiratory disease.
6. Severe renal or hepatic impairment.
7. Allergy to drugs used in the study.
8. Known substance abuse.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
The change in the degree of postoperative pain | 0, 3, 6, 12, 24, 36 and 48 hours; where T0= time of arrival of the patient to PACU.
  The change in the degree of pain will be evaluated using according to visual analogue scale (VAS) where 0= no pain, and 10= worst pain possible. If VAS is ≥4= inadequate pain relief,

CONTACTS AND LOCATIONS:
Overall Officials: Salwa H Waly, Principal Investigator — Faculty of medicine. Zagazig University. Egypt
Locations (1):
- Zagazig Univesity, Zagazig, Sharqia Province, Egypt